CLINICAL TRIAL: NCT02715063
Title: High Intensity Interval- vs Resistance or Combined- Training for Improving Cardiometabolic Health in Overweight Adults (Cardiometabolic HIIT-RT Study): Study Protocol for a Factorial Randomised Controlled Trial
Brief Title: Cardiometabolic HIIT-RT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas (Other)
Collaborators: Universidad del Rosario (Other); Universidad Manuela Beltrán (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 06-1006-2014
Record Dates: First submitted 2016-03-08; First posted 2016-03-22 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Metabolic Diseases; Overweight; Motor Activity
MeSH Terms: conditions — Metabolic Diseases; Overweight; Motor Activity | interventions — High-Intensity Interval Training; Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Intensity Interval (Experimental): Walking on a treadmill 4min at 80-90% peak heart rate and recovery 4 min at 65% peak heart rate until expenditure of 300 kcal during adaptation (first 4 weeks) and 500 kcal after week number 4 until the end of training.
  Interventions: Behavioral: High Intensity Interval
- Resistance training (Active Comparator): Completing a resistance circuit (including upper and lower muscle groups) as many times as needed according to subject weight until expenditure of 300 kcal during adaptation (first 4 weeks) at 20-30% of 1 one-rep max and 500 kcal after week number 4 until the end of training, at 40-60% of one-rep max.
  Interventions: Behavioral: Resistance training
- Plus: High Intensity Interval + Resistance Training (Active Comparator): Walking on a treadmill as intervention 1 until 50% the energy expenditure prescribed is reached, then completing a resistance circuit until 100% energy expenditure is reached. Exercise will be performed at three sessions per week.
  Interventions: Behavioral: Plus: High Intensity Interval + Resistance Training
- Usual clinical care (Placebo Comparator): This group will receive the usual clinical care according to the consensus recommendations of the national goals for cardiovascular health promotion and disease reduction of the American Heart Association and Colombian guidelines COLDEPORTES.
  Interventions: Other: Usual clinical care

INTERVENTIONS:
Behavioral: High Intensity Interval — Exercise will be performed at three sessions per week. All sessions will be supervised by a trained health or exercise professional.
  Arms: High Intensity Interval
Behavioral: Resistance training — Exercise will be performed at three sessions per week. All sessions will be supervised by a trained health or exercise professional.
  Arms: Resistance training
Behavioral: Plus: High Intensity Interval + Resistance Training — Exercise will be performed at three sessions per week. All sessions will be supervised by a trained health or exercise professional.
  Arms: Plus: High Intensity Interval + Resistance Training
Other: Usual clinical care — Dietary restriction (1300-1500kcal) 50-52% carbohydrates, 33-35% fat, 15-20% protein
  Arms: Usual clinical care

SUMMARY:
Several studies have shown relationship between exercise intensity and improvement cardiometabolic health such as body composition, endothelial function, blood pressure and blood lipids. It has been suggested that high intensity interval training and also strength or resistance training generate positive effects on metabolic risk factors, nevertheless the comparison between both types of training and their combination has not yet provided conclusive evidence. Also, it has been shown that dietary restriction has similar or more positive effects that exercise alone and the effect is greater when it is combined with exercise. For these reasons, it is necessary to clarify which type of training, in combination with a dietary restriction, is more effective to improve cardiometabolic health

DETAILED DESCRIPTION:
The investigators hypothesized that high intensity interval, resistance training or combined training would result in similar improvements in cardiometabolic health as compared to the usual clinical care in a cohort of sedentary overweight (age 30-50 years old).

ELIGIBILITY:
Inclusion Criteria:

* Meets at least one criteria for metabolic Syndrome (IDF 2006): Central obesity: waist circumference ≥90cm (men) ≥80cm (women); triglycerides ≥ 150mg/dl; HDL-c <40mg/dl (men) <50 (women); Blood pressure ≥130/85mmHg and fasting plasma glucose ≥ 100mg/dL.
* Written informed consent.
* Interested in improving health and fitness.

Exclusion Criteria:

* Systemic infections.
* Weight loss or gain of >10% of body weight in the past 6 months for any reason.
* Currently taking medication that suppresses or stimulates appetite.
* Uncontrolled hypertension: systolic blood pressure 160 mm Hg or diastolic blood pressure 95 mm Hg on treatment.
* Gastrointestinal disease, including self-reported chronic hepatitis or cirrhosis, any episode of alcoholic hepatitis or alcoholic pancreatitis within past year, inflammatory bowel disease requiring treatment in the past year, recent or significant abdominal surgery (e.g., gastrectomy).
* Asthma.
* Diagnosed diabetes (type 1 or 2), fasting impaired glucose tolerance (blood glucose 118 mg/dL), or use of any anti-diabetic medications.
* Currently taking antidepressant, steroid, or thyroid medication, unless dosage is stable (no change for 6 months).
* Any active use of illegal or illicit drugs.
* Current exerciser (>30 min organized exercise per week).
* Indication of unsuitability of current health for exercise protocol (PARQ).
* Any other conditions which, in opinion of the investigators, would adversely affect the conduct of the trial.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in endothelial function as measured by flow-mediated vasodilation (FMD) | Baseline and 12 weeks immediately after the interventions ends
  FMD will be measured using the guidelines reported by Corretti et al. The diameter of the brachial artery will be assessed using a high-resolution ultrasound device (Siemens SG-60, USA), equipped with a 7.5 MHz linear array transducer.

SECONDARY OUTCOMES:
Change from Baseline in body Composition as measured by Dual Energy X-ray Absorptiometry | Baseline and 12 weeks immediately after the interventions ends
  Changes in abdominal and total adiposity (DEXA), lean tissue mass and bone mass (DEXA) the 12 weeks intervention program
Body Weight | Baseline and 12 weeks immediately after the interventions ends
Body Mass Index | Baseline and 12 weeks immediately after the interventions ends
  BMI will be calculated as the body weight in kilograms divided by the square of the height in meters.
Blood Pressure | Baseline and 12 weeks immediately after the interventions ends
Change from Baseline in peak uptake of volume of oxygen | Baseline and 12 weeks immediately after the interventions ends
  It will be determined using a maximum treadmill exercise test (Precor TRM 885, Italy) following the modified Balke protocol
Change from Baseline in muscular fitness | Baseline and 12 weeks immediately after the interventions ends
  Muscular fitness (MF) will be assessed using handgrip test (maximum handgrip strength assessment) using a standard adjustable handle analogue handgrip dynamometer T-18 TKK SMEDLY III®
Change from Baseline in Flexibility using the sit and reach test | Baseline and 12 weeks immediately after the interventions ends
Change from Baseline in LDL Cholesterol | Baseline and 12 weeks immediately after the interventions ends
Change from Baseline in HDL Cholesterol | Baseline and 12 weeks immediately after the interventions ends
Change from Baseline in Triglycerides | Baseline and 12 weeks immediately after the interventions ends
Change from Baseline in Glucose | Baseline and 12 weeks immediately after the interventions ends
Change from Baseline in Hemoglobin A1c | Baseline and 12 weeks immediately after the interventions ends
Change from Baseline in Quality & satisfaction with life by SF Community - short-form survey (SF-12™) Colombian version | Baseline and 12 weeks immediately after the interventions ends
Change from Baseline in Heart rate variability | Baseline and 12 weeks immediately after the interventions ends
  HRV will be performed according to current recommendations by European Society of Cardiology using an evaluated share-ware
24-hour dietary recall | Baseline and 12 weeks immediately after the interventions ends
  Dietary data will be collected from participants on 24h of their study enrollment. Prior to administration of the 24HR, each subject received two-dimensional food models with depiction of foods and serving sizes in order to assist in reporting portion sizes of food intake.
Aortic pulse wave velocity (PWVao) and augmentation index (AIx) | Baseline and 12 weeks immediately after the interventions ends
  PWVao and AIx will be measured with oscillometric method using the occlusion technique.

CONTACTS AND LOCATIONS:
Overall Officials: Robinson Ramírez Vélez, Ph.D, Principal Investigator — Universidad del Rosario
Locations (1):
- Robinson Ramírez Vélez Ph.D, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez-Velez R, Correa-Bautista JE, Gonzalez-Ruiz K, Tordecilla-Sanders A, Garcia-Hermoso A, Schmidt-RioValle J, Gonzalez-Jimenez E. The Role of Body Adiposity Index in Determining Body Fat Percentage in Colombian Adults with Overweight or Obesity. Int J Environ Res Public Health. 2017 Sep 21;14(10):1093. doi: 10.3390/ijerph14101093. PMID 28934175
- [Derived] Ramirez-Velez R, Hernandez A, Castro K, Tordecilla-Sanders A, Gonzalez-Ruiz K, Correa-Bautista JE, Izquierdo M, Garcia-Hermoso A. High Intensity Interval- vs Resistance or Combined- Training for Improving Cardiometabolic Health in Overweight Adults (Cardiometabolic HIIT-RT Study): study protocol for a randomised controlled trial. Trials. 2016 Jun 24;17(1):298. doi: 10.1186/s13063-016-1422-1. PMID 27342073